CLINICAL TRIAL: NCT02277704
Title: A Phase 2, Double-Blind, Randomized, Multicenter, Placebo-Controlled Study to Evaluate the Efficacy and Safety of TNX-102 SL Taken at Bedtime in Subjects With Military-Related PTSD and Related Conditions (Protocol No. TNX-CY-P201) -"AtEase STUDY"
Brief Title: Safety and Efficacy Study of TNX-102 SL in Subjects With Military-Related PTSD and Related Conditions
Acronym: AtEase
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tonix Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TNX-CY-P201
Record Dates: First submitted 2014-10-23; First posted 2014-10-29 (Estimated); Results first posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-05

CONDITIONS: PTSD
Keywords: PTSD; Military-related PTSD and other related conditions
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): 2 x placebo tablet ("placebo") to be taken sublingually once daily at bedtime.
  Interventions: Drug: Placebo
- TNX-102 SL, 2.8 mg (Active Comparator): 1 x TNX-102 SL 2.8mg tablet ("TNX-102 SL") and 1 x placebo tablet ("placebo") to be taken sublingually once daily at bedtime.
  Interventions: Drug: TNX-102 SL; Drug: Placebo
- TNX-102 SL, 5.6 mg (Active Comparator): 2 x TNX-102 SL 2.8mg tablets ("TNX-102 SL") to be taken sublingually once daily at bedtime.
  Interventions: Drug: TNX-102 SL

INTERVENTIONS:
Drug: TNX-102 SL
  Arms: TNX-102 SL, 2.8 mg; TNX-102 SL, 5.6 mg
Drug: Placebo
  Arms: Placebo; TNX-102 SL, 2.8 mg

SUMMARY:
This is a 12-week, multicenter, randomized, double-blind, placebo-controlled, fixed-dose, parallel-group study that will investigate the efficacy and safety of two doses of TNX-102 SL -a sublingual formulation of cyclobenzaprine. Following successful screening and randomization, eligible subjects will return regularly to the study clinic for weekly or biweekly visits for assessments of efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 65 years of age
* Diagnosed with current PTSD as defined by the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5),
* For patients with a qualifying Index trauma(s) resulting in PTSD that occurred during military service, military contractor, Department of Homeland Security or law enforcement
* Willing and able to withdraw and refrain from specific therapies (ask PI)
* Use medically acceptable form of contraception (female only)
* Signed informed consent

Exclusion Criteria:

* Significant traumatic brain injury
* Severe depression
* Bipolar and psychotic disorders
* Increase risk of suicide
* Significant clinical (cardiac, systemic infection, drug/alcohol abuse) or laboratory abnormalities (including positivity for Hep B, Hep C, HIV)
* Unable to wash-out specific medications (ask PI)
* History of violent behavior within past 2 years, unrelated to work duties
* History of drug or alcohol abuse within past 6 months
* Positive illegal substance test
* Known hypersensitivity to cyclobenzaprine
* Others: seizure disorders, uncontrolled sleep apnea, BMI>40
* Participation in an investigational study in past 30 days
* In the process of litigating for compensation for a psychiatric disorder
* Females that are pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise Bedoya, Study Director — Premier Research
Locations (23):
- United States (23):
  - Tuscaloosa VA Medical Center, Tuscaloosa, Alabama
  - Noesis Pharma, Phoenix, Arizona
  - Sun Valley Research Center, Imperial, California
  - National City, National City, California
  - Excell Research, Inc, Oceanside, California
  - Neuropsychiatric Research Center of Orange County, Orange, California
  - CITRIALS, Riverside, California
  - Veteran Affairs, San Diego Health Care System, San Diego, California
  - Cns, Inc., Torrance, California
  - Sarkis Clinical Trials, Lake City, Florida
  - Compass Research North, LLC, Leesburg, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Atlanta Center For Medical Research, Atlanta, Georgia
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Novex Clinical Research, New Bedford, Massachusetts
  - Premier Psychiatric Research Institute, Inc., Lincoln, Nebraska
  - Altea Research, Las Vegas, Nevada
  - Cedarhurst, Cedarhurst, New York
  - Cincinnati, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Clinical Trials of Texas, San Antonio, Texas
  - Northwest Clinical Research Center, Bellevue, Washington

REFERENCES:
- [Result] Sullivan GM, Gendreau RM, Gendreau J, Peters P, Peters A, Engels J, Daugherty BL, Vaughn B, Weathers FW, Lederman S. Randomized clinical trial of bedtime sublingual cyclobenzaprine (TNX-102 SL) in military-related PTSD and the role of sleep quality in treatment response. Psychiatry Res. 2021 Jul;301:113974. doi: 10.1016/j.psychres.2021.113974. Epub 2021 Apr 30. PMID 33979763

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: 2 x placebo tablet ("placebo") to be taken sublingually once daily at bedtime.
  Placebo
- TNX-102 SL, 2.8 mg: 1 x TNX-102 SL 2.8mg tablet ("TNX-102 SL") and 1 x placebo tablet ("placebo") to be taken sublingually once daily at bedtime.
  TNX-102 SL
  Placebo
- TNX-102 SL, 5.6 mg: 2 x TNX-102 SL 2.8mg tablets ("TNX-102 SL") to be taken sublingually once daily at bedtime.
  TNX-102 SL
Period: Overall Study
Arm/Group | Placebo | TNX-102 SL, 2.8 mg | TNX-102 SL, 5.6 mg
Started | 94 | 101 | 50
Completed | 67 | 71 | 41
Not Completed | 27 | 30 | 9

BASELINE CHARACTERISTICS:
Groups:
- TNX-102 SL, 2.8 mg: 1 x TNX-102 SL 2.8 mg tablet ("TNX-102 SL") and 1 x placebo tablet ("placebo") to be taken sublingually once daily at bedtime.
- Total: Total of all reporting groups
Arm/Group | Placebo | TNX-102 SL, 2.8 mg | TNX-102 SL, 5.6 mg | Total
Number analyzed (Participants) | 94 | 101 | 50 | 245
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 31.9 (6.48) | 34.5 (8.11) | 34.7 (8.93) | 33.6 (7.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 4 | 19
  Male | 88 | 92 | 46 | 226
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 15 | 11 | 46
  Not Hispanic or Latino | 74 | 86 | 39 | 199
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 0 | 4
  Asian | 3 | 1 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 21 | 27 | 12 | 60
  White | 61 | 68 | 33 | 162
  More than one race | 4 | 1 | 0 | 5
  Unknown or Not Reported | 4 | 1 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: The Mean Change From Baseline (Visit 2) in the Total CAPS-5 Score After 12 Weeks of Treatment Evaluated at Visit 9 (Week 12).
Description: The mean change from baseline (Visit 2) in the Total CAPS-5 score after 12 weeks of treatment evaluated at Visit 9 (Week 12). The primary efficacy comparison will be the change from baseline in total CAPS-5 score for the 2.8 mg treatment arm compared to placebo. CAPS-5 score ranges from 0-80 with lower scores indicating less severe PTSD symptoms.
Time Frame: Day 1, Week 12
Population: Results are reported for patients in mITT population (included all patients who were randomized, had a baseline CAPS-5 and at least one post-baseline CAPS-5).
  At Week 12 or last visit for subjects discontinuing early, values recorded more than 7 days after the last recorded dose are censored. Subjects that are lost to follow up or do not have a last dose date recorded have the day before their final visit imputed as the last dose date.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | TNX-102 SL, 2.8 mg | TNX-102 SL, 5.6 mg
Number analyzed (Participants) | 92 | 90 | 49
units on a scale | -17.0 (1.98) | -19.2 (1.99) | -21.5 (2.41)

2. Secondary Outcome: Change From Baseline in Patients' Quality of Sleep Using the PROMIS Sleep Disturbance Scale After 12 Weeks of Treatment
Description: Change from baseline in patients' quality of sleep using the PROMIS (Patient -Reported Outcome Measurement Information System) Sleep Disturbance scale after 12 weeks of treatment comparing the 2.8 mg treatment arm to placebo. Raw scores are converted to T-scores using published conversion tables. Sleep Disturbance T-score ranges from 28.9 to 76.5. Lower scores indicate less sleep disturbance
Time Frame: Day 1, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | TNX-102 SL, 2.8 mg | TNX-102 SL, 5.6 mg
Number analyzed (Participants) | 92 | 90 | 49
units on a scale | -7.9 (1.72) | -11.1 (1.74) | -11.0 (2.10)

3. Secondary Outcome: Clinician Global Impression - Improvement Scale Responder Rate at Week 12
Description: Responder rates in CGI-I (Clinician Global Impression - Improvement Scale) after 12 weeks of treatment comparing the 2.8 mg treatment arm to placebo. Responder rate is defined as the number of patients scored as either a 1 or 2 on CGI-I at Week 12. The score ranges from 1 to 7 with the following anchors for each score:1=Very much improved, 2=Much improved, 3=Minimally improved, 4=No change, 5=Minimally worse, 6=Much worse, 7=Very much worse
Time Frame: Week 12
Population: Results are reported for patients in mITT population (included all patients who were randomized, had a baseline CAPS-5 and at least one post-baseline CAPS-5). Patients without CGI-I data at Week 12 were considered as being non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TNX-102 SL, 2.8 mg | TNX-102 SL, 5.6 mg
Number analyzed (Participants) | 92 | 90 | 49
Participants | 41 | 48 | 31

4. Secondary Outcome: Mean Change From Baseline in Sheehan Disability Scale (SDS) Total Score
Description: Mean Change from Baseline in SDS Total Score at Week 12. Score ranges from 0 to 30. A score of 0 means the patient is unimpaired, and a score of 30 means the patient is highly impaired.
Time Frame: Day 1, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | TNX-102 SL, 2.8 mg | TNX-102 SL, 5.6 mg
Number analyzed (Participants) | 92 | 90 | 49
units on a scale | -6.4 (1.11) | -7.9 (1.11) | -8.7 (1.35)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: All adverse events are reported for the Safety Population, which includes patients who took at least one dose of study medication.
  All-cause mortality is reported for all patients.
Arm/Group | Placebo | TNX-102 SL, 2.8 mg | TNX-102 SL, 5.6 mg
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/101 | 0/50
Serious Adverse Events (participants affected / at risk) | 3/94 | 0/93 | 1/50
Other Adverse Events (participants affected / at risk) | 36/94 | 59/93 | 35/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=94) | TNX-102 SL, 2.8 mg (N=93) | TNX-102 SL, 5.6 mg (N=50)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Perirectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — acute episode of multiple sclerosis
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=94) | TNX-102 SL, 2.8 mg (N=93) | TNX-102 SL, 5.6 mg (N=50)
Hypoaesthesia Oral (Gastrointestinal disorders) | 2 | 36 | 18
Dry mouth (Gastrointestinal disorders) | 10 | 4 | 8
paraesthesia oral (Gastrointestinal disorders) | 3 | 15 | 2
Glossodynia (Gastrointestinal disorders) | 1 | 3 | 3
Somnolence (Nervous system disorders) | 6 | 11 | 8
Headache (Nervous system disorders) | 4 | 5 | 6
Sedation (Nervous system disorders) | 1 | 2 | 6
Insomnia (Psychiatric disorders) | 8 | 7 | 3
Abnormal dreams (Psychiatric disorders) | 5 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 3 | 2
Weight Increased (Investigations) | 5 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An industry standard NDA is in place with all investigators.